CLINICAL TRIAL: NCT05838690
Title: Optimizing Tracheal Intubation Outcomes and Neonatal Safety
Acronym: OPTION SAFE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 22-019975; R01HD106996 (NIH)
Record Dates: First submitted 2023-03-14; First posted 2023-05-01 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Infant; Intubation Complication
Keywords: Infant; Intubation; NICU; Safety

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-Intervention Phase (No Intervention): NICU Patients who are intubated without the PINS Bundle.
- Post-intervention Phase (Active Comparator): NICU Patients who are intubated after unit implementation of the PINS Bundle
  Interventions: Other: Personalized Intubation Safety (PINS) Bundle

INTERVENTIONS:
Other: Personalized Intubation Safety (PINS) Bundle — The Personalized Intubation Safety (PINS) Bundle addresses 5 core domains that are individualized to the patient to develop a prospective, personalized and comprehensive multidisciplinary intubation plan: (1) patient risk assessment; (2) treatment threshold for intubation; (3) premedication (promoting paralytic premedication); (4) equipment (promoting video laryngoscope); (5) provider selection and escalation plan
  Other Names: PINS Bundle
  Arms: Post-intervention Phase

SUMMARY:
The purpose of the study is to assess the impact of a personalized intubation planning tool, the Personalized INtubation Safety (PINS) Bundle on intubation procedural safety and clinical outcomes among patients intubated in the neonatal intensive care unit (NICU) setting.

DETAILED DESCRIPTION:
Tracheal intubation (TI) in the neonatal intensive care unit (NICU) is frequently complicated by adverse safety outcomes such as adverse tracheal intubation associated events, multiple TI attempts, and oxygen desaturation. Investigators have developed, refined, and tested a Personalized INtubation Safety (PINS) Bundle that targets a prospective and individualized approach to TI planning and management. The Prospective Intubation Safety (PINS) Bundle addresses 5 core evidence-based domains that are individualized to the patient to develop a prospective, personalized and comprehensive multidisciplinary TI plan: (1) patient risk assessment; (2) treatment threshold for intubation; (3) premedication (promoting paralytic medication); (4) equipment (promoting video laryngoscope); (5) provider selection and escalation plan.

This is a pragmatic stepped wedge cluster randomized trial of NICU patients who are intubated across 8 participating hospitals to determine if the PINS Bundle, compared to no PINS Bundle, reduces the incidence of adverse tracheal intubation associated events.

The primary objective of this study is to determine the effectiveness of the PINS Bundle to decrease adverse TI safety events. The secondary objectives are 1) to evaluate if the impact of the PINS Bundle on adverse TI safety events varies based on provider skill, and 2) to determine the impact of the PINS Bundle on NICU clinical outcomes of extubation failure, duration of intubation, NICU mortality, and intraventricular hemorrhage.

ELIGIBILITY:
Inclusion Criteria:

Infants undergoing tracheal intubation in the neonatal intensive care unit (NICU)

Exclusion Criteria:

Endotracheal tube exchanges, as this represents a distinct procedure.

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3000 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Tracheal intubation associated event (TIAE) | During the intubation procedure, on average 20 minutes
  Any adverse tracheal intubation associated event (TIAE) during the intubation encounter. In NEAR4NEOS database, a comprehensive group of adverse TIAEs are based on standard consensus-based definitions and classified as severe and non-severe

SECONDARY OUTCOMES:
Severe TIAE | During the intubation procedure, on average 20 minutes
  Any severe TIAE, defined by National Emergency Airway Registry for Neonates (NEAR4NEOS) Operational Definitions
Magnitude of oxygen desaturation | During the intubation procedure, on average 20 minutes
  Difference between highest oxygen saturation (SpO2) value immediately before first intubation attempt and lowest value at any point during the procedure
Number of subjects with multiple intubation attempts (>2 attempts) | During the intubation procedure, on average 20 minutes
  More than 2 intubation attempts
Duration of mechanical ventilation | Through study completion, on average 90 days
  Duration of mechanical ventilation after the immediate intubation encounter
Number of subjects requiring reintubation within 24 hours of extubation | Up to 24 hours after extubation
  Need for reintubation within 24 hours of extubation from the course of ventilation immediately following the intubation encounter
Number of subjects with Intraventricular hemorrhage | Up to 7 days after birth
  Any intraventricular hemorrhage and grade on head ultrasound, assessed for at risk preterm infants
NICU Mortality | Through study completion, on average 90 days
  Death before NICU discharge

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Foglia, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (8):
- United States (7):
  - University of Arkansas Medical Sciences, Little Rock, Arkansas
  - University of Colorado - Denver, Denver, Colorado
  - Yale-New Haven Hospital, New Haven, Connecticut
  - Dartmouth-Hitchcock Clinic, Lebanon, New Hampshire
  - WakeMed Health & Hospitals, Raleigh, North Carolina
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - University of Washington, Seattle, Washington
- CHU Sainte-Justine, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
The PI will share unique research resources developed through this NIH-funded grant to enhance the value and further the advancement of research. The PI will make data available after study completion and in accordance with NIH policies. The data will only be provided to those investigators who agree to adhere to a signed research data use agreement. The execution of the agreement will require approval by the Children's Hospital of Philadelphia (CHOP) Institutional Review Board (IRB) or demonstration of IRB exemption per institutional policy. The data and associated documentation will be available to users only under a data-sharing agreement that provides for: (1) a commitment to using the data only for research purposes and does not identify any individual participant; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying or returning the data after analyses are completed
Time Frame: Data will be available after study completion
Access Criteria: The data and associated documentation will be available to users only under a data-sharing agreement that provides for: (1) a commitment to using the data only for research purposes and does not identify any individual participant; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying or returning the data after analyses are completed